CLINICAL TRIAL: NCT02459028
Title: A Phase II, Community-based, Single-blinded, Randomized Controlled, Parallel-group Trial to Assess the Effects of a Tailored Positive Psychology Intervention on Chronic Pain and Well-being in Individuals With Spinal Cord Injury
Brief Title: Positive Psychology Interventions in Individuals With Chronic Pain and Spinal Cord Injury
Acronym: T3P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-24
Record Dates: First submitted 2015-02-16; First posted 2015-06-01 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Spinal Cord Injury
MeSH Terms: conditions — Chronic Pain; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- T3P Intervention group (Experimental): Intervention group: Participants are instructed to practice 4 out of 10 different Positive Psychology Exercises (Gratitude, Optimism, Act of Kindness, Social Relations, Forgiveness, Flow, Savoring, Goals, Spirituality, Taking Care of the Body) for at least 15 minutes, at least one day every week including on "bad" days (defined as days with higher than average levels of pain intensity or feeling "down in the dumps") for 8 weeks.
  Interventions: Behavioral: Positive Psychology intervention
- Control group (Active Comparator): Control group: Control Exercise (Attention Training): Participants assigned to the control group are instructed to be more attentive to their surroundings and write about three specific events or activities from the past 7 days for at least 15 minutes once a week for 8 weeks. This condition is designed to control for the effects of time and participation in an intervention activity.
  Interventions: Behavioral: Positive Psychology intervention (Control exercise)

INTERVENTIONS:
Behavioral: Positive Psychology intervention — Intervention group: Participants are instructed to practice 4 out of 10 differentPositive Psychology Exercises (Gratitude, Optimism, Act of Kindness, Social Relations, Forgiveness, Flow, Savoring, Goals, Spirituality, Taking Care of the Body) for at least 15 minutes, at least one day every week including on "bad" days (defined as days with higher than average levels of pain intensity or feeling "down in the dumps") for 8 weeks.
  Arms: T3P Intervention group
Behavioral: Positive Psychology intervention (Control exercise) — Control group: Control Exercise (Attention Training): Participants assigned to the control group are instructed to be more attentive to their surroundings and write about three specific events or activities from the past 7 days for at least 15 minutes once a week for 8 weeks. This condition is designed to control for the effects of time and participation in an intervention activity.
  Arms: Control group

SUMMARY:
Background:

Chronic pain is one of the most burdensome potential consequences of a physical disability, such as spinal cord injury (SCI). Estimates of the incidence of chronic pain in SCI range between 65 - 80%. A recent pilot-study of a computer-based tailored positive psychology intervention showed a significant reduction in pain intensity, pain interference, pain catastrophizing and depression and an enhancement of subjective well-being and control over pain in persons with chronic pain secondary to a physical disability.

Study Objective:

Objective 1: To determine the efficacy of a tailored positive psychology intervention (T3P) in a community-based, single-blind, randomized, controlled, parallel group trial on subjective well-being and pain in individuals with chronic pain secondary to SCI.

Hypothesis 1: T3P will result in (1) greater immediate and long-lasting increase in subjective well-being, and perceived control over pain and (2) greater immediate and long-lasting decrease in depression, pain intensity, pain interference and catastrophizing, relative to an active control treatment.

Specific aim 1: To increase the understanding of the mechanisms underlying T3P by determining potential mediation effects.

Hypothesis 2: (1) Pain catastrophizing and pain control mediate the effect of T3P on pain intensity, and (2) positive and negative affect mediate the effect of T3P on life satisfaction and depression.

Objective 2: To identify for whom T3P is most effective by exploring potential moderator effects.

Study Design:

The proposed study is a single-blind, randomized, controlled trial with a parallel group design to determine the effects and mechanisms of T3P in a Swiss community sample of persons with chronic pain secondary to SCI.

ELIGIBILITY:
Inclusion Criteria:

* Registered in Swiss Spinal Cord Injury Cohort Study (SwiSCI)
* Individuals who experience an average disability-related pain intensity of ≥ 4 on a 0-10 numeric rating scale in the past week
* Individuals who experience pain at least half the days in the past four weeks, and
* Individuals are able to speak, read and write German

Exclusion Criteria:

* Individuals who report current participation in any psychotherapy (e.g. psychotherapy, hypnosis, biofeedback) once a month or more often
* Individuals who report hospitalization for psychiatric reasons within the past year
* Individuals with a severe cognitive impairment defined as one or more errors on a Six-Item Screening

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain Numeric Rating Scale (pain intensity) | Baseline (Pre-treatment)
  Pain Numeric Rating Scale (0-10)
Change from baseline in Pain Numeric Rating Scale (pain intensity) at Mid-treatment | Mid-treatment (at 4 weeks)
  Pain Numeric Rating Scale (0-10)
Change from baseline in Pain Numeric Rating Scale (pain intensity) at Post-treatment | Post-treatment (at 8 weeks)
  Pain Numeric Rating Scale (0-10)
Change from baseline in Pain Numeric Rating Scale (pain intensity) at Follow-up | Follow-up (at 20 weeks or at 3 months after post-treatment)
  Pain Numeric Rating Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Müller, Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic Research, Nottwil, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Muller R, Segerer W, Ronca E, Gemperli A, Stirnimann D, Scheel-Sailer A, Jensen MP. Inducing positive emotions to reduce chronic pain: a randomized controlled trial of positive psychology exercises. Disabil Rehabil. 2022 Jun;44(12):2691-2704. doi: 10.1080/09638288.2020.1850888. Epub 2020 Dec 2. PMID 33264568